CLINICAL TRIAL: NCT02416856
Title: Brain Connectivity Supporting Language Recovery in Aphasia
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: R01-Bonilha; R01DC014021 (NIH)
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Aphasia; Stroke; Speech Disorders; Communications Disorders
Keywords: Aphasia; Brain; Stimulation; Communication; Stroke; Speech Disorders; Communications Disorders; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms
MeSH Terms: conditions — Aphasia; Stroke; Speech Disorders; Communication Disorders; Communication; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The integrity of structural connectivity supporting cortical regions in the left brain hemisphere is hypothesized to enable treatment-induced naming recovery in persons with language difficulties after a stroke (aphasia). The investigators will map whole brain connectivity (i.e., the brain connectome) to investigate the role of cortical connectivity in impairment (Aim 1) and recovery (Aim 2) in patients with aphasia undergoing treatment. This information will be used to construct personalized markers of anomia treatment outcome (Aim 3), which may serve as a guide for speech-language pathologists and neurologists when facing patient management decisions.

DETAILED DESCRIPTION:
Aphasia, an impairment of language processing, is one of the most common consequences of strokes affecting the dominant brain hemisphere4. Patients with aphasia are usually incapable of working, and their interactions with family and friends are often severely affected. The hallmark deficit of aphasia is the inability to name objects or people (anomia)12. The severity of anomia is closely related to a poor quality of life.

While many patients with aphasia exhibit some language recovery in the first days to weeks after the stroke, 30-40% persist with long lasting naming impairments4. Fortunately, speech therapy can be very effective to improve naming for some patients with chronic aphasia5-8. However, it is well recognized among clinicians that speech therapy can be ineffective for other patients, making it difficult to predict how and why some patients benefit from naming treatment, while others show little or no improvement.

Here, the investigators propose to evaluate whether naming impairment and naming recovery are related to the extent of structural damage to the cortical language network. Importantly, the investigators will evaluate damage as the combined effect of cortical necrosis and cortical disconnection. The investigators hypothesize that assessing anomia as being either due to gray matter necrosis or due to cortical disconnection constitutes a false dichotomy since most chronic patients exhibit gray and white matter damage. Furthermore, the investigators propose that disconnection of seemingly spared cortical areas has up till now been underappreciated in patients with stroke due to limitations in brain connectivity assessment tools. By examining only areas of cortical necrosis without considering disconnected areas, one may underestimate the magnitude of language network damage. A better understanding of the effects from both cortical damage and disconnection on anomia and its recovery could lead to an improved clinical management of aphasia.

The investigators will employ the innovative concept of the brain connectome, i.e., the individualized map of neural connections in the brain, to evaluate whether naming recovery is supported by preserved gray matter and preserved connectivity involving key language areas in the left hemisphere. The investigators propose that left frontal and left temporal connectivity mapped based on the individual's connectome is an important explanatory variable towards naming impairment and recovery.

The investigators believe that this research is significant for the three main reasons. First, it can have a direct clinical impact by providing a better understanding of which patients can benefit from therapy. Second, it can unveil the neurobiological mechanisms supporting language recovery, improving our understanding of brain plasticity related to language rehabilitation. Finally, if disconnection contributes to language impairment, our methods can be developed to test specific theories of language organization in the brain. The significance of these aspects is explained in detail below.

ELIGIBILITY:
Criteria:No new patients will be recruited for the current project. We will rely solely on data collection in the tDCS-Trial (U01 DC011739, period 7/1/2012-6/31/2017).

Following is the Eligibility for the TDCS-Trial:

Inclusion Criteria:

1. Patients must be willing and able to give informed consent.
2. Patients must be willing and able to comply with study requirements.
3. Patients must be between 25- and 80-years of age.
4. Patients must be native English speakers.
5. Patients must be pre-morbidly right-handed.
6. Patients must have sustained a one-time ischemic stroke in the left-hemisphere.
7. Patients must be greater than 6-months post-stroke.
8. Patients must have an aphasia diagnosis as confirmed by the Western Aphasia Battery-Revised.
9. Patients must be MRI-compatible (e.g., no metal implants, not claustrophobic, etc.).
10. Patients must achieve at least 65% accuracy on naming task during screening -

Exclusion Criteria:

1. History of brain surgery
2. Seizures during the previous 12 months
3. Sensitive scalp (per patient report)
4. Able to overtly name more than an average of 140 out of 175 items during the pre-treatment picture naming test (Philadelphia Naming Test) during Visits 2 or 3.
5. Unable to overtly name at least an average of 5 out of 80 items during the pre-treatment fMRI sessions during Visits 2 or 3.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No new patients will be recruited for the current project. We will rely solely on data collection in the tDCS-Trial (U01 DC011739, period 7/1/2012-6/31/2017). All information used in our experiments will be available as a result of the standardized set of tests that patients undergo in the trial.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Improvement in naming performance as assessed by the number of correctly spoken words after therapy | 5 years
  The primary outcome measure of this study is the objective improvement in the number of correctly spoken words after therapy. This study is also aimed at evaluating the neurological mechanisms (i.e., integrity of brain networks after stroke) that enable therapy-induced improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo F Bonilha, MD, Principal Investigator — Assistant Professor
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States